CLINICAL TRIAL: NCT02748785
Title: Effect of Methotrexate Discontinuation on Efficacy of Seasonal Influenza Vaccination in Patients With Rheumatoid Arthritis: A Randomized Clinical Trial
Brief Title: MTX Discontinuation and Vaccine Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-IMJ-001
Record Dates: First submitted 2015-09-08; First posted 2016-04-22 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2017-11

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (No MTX Hold before Vaccination) (Experimental): Group 1 will continue MTX
  Interventions: Drug: Methotrexate; Biological: Seasonal Influenza vaccine
- Group 2 (MTX hold 4 Weeks before vaccination) (Experimental): Group 2 will hold MTX 4 weeks before vaccination and resume MTX on the day of vaccination
  Interventions: Drug: Methotrexate; Biological: Seasonal Influenza vaccine
- Group 3 (MTX hold 2 Weeks before Vaccination) (Experimental): Group 3 will hold MTX 2 weeks before vaccination and resume MTX 2 weeks after vaccination
  Interventions: Drug: Methotrexate; Biological: Seasonal Influenza vaccine
- Group 4 (MTX hold on Day of Vaccination) (Experimental): Group 4 will hold MTX on day of vaccination and resume MTX 4 weeks after vaccination.
  Interventions: Drug: Methotrexate; Biological: Seasonal Influenza vaccine

INTERVENTIONS:
Drug: Methotrexate — Methotrexate will be continued
Biological: Seasonal Influenza vaccine — all subjects will be vaccinated with a seasonal influenza vaccine

SUMMARY:
To investigate whether a short term discontinuation of methotrexate (MTX) will improve the vaccination efficacy to seasonal influenza vaccination without deteriorating RA disease activity in a randomized clinical trial.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic inflammatory disease that affects the joints as the main target of the inflammation. Patients with RA require chronic treatment with disease modifying anti-rheumatic drugs (DMARDs) including methotrexate (MTX), which constitutes the mainstay of treatment.

Underlying immune dysfunction and the additional immune suppression associated with treatment render patients with RA more susceptible to infection. Thus, vaccination against preventable diseases including influenza, pneumococcal pneumonia and hepatitis B is recommended for all RA patients who are subject to treatment with immunesupprssive drugs, unless there is a contraindication to the use of vaccination. However, low dose of glucocorticoids, conventional DMARDs and biological DMARDs including tumor necrosis factor inhibitors have been reported to substantially decrease vaccine response (4); MTX has been reported to be associated with a decreased response to seasonal influenza vaccination by up to 15%.

To optimize a vaccine response, vaccination should be administrated before the treatment with immunesuppressive medications is initiated. However, most patients with RA are already on stable dose of DMARDs at the time of when vaccinations, especially vaccine against seasonal influenza that needs annual administration, are considered. Alternatively, temporarily discontinuation of DMARDs might restore normal immune response to and so improve the efficacy of vaccination.

Although a short term discontinuation of DMARDs during perioperative period has not been associated with increased disease activity the longer discontinuation of DMARDs might lead to a significant aggravation of RA disease activity. To optimize the vaccine response, a short term discontinuation of DMARDs could be considered if this approach proves to be safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 years at time of consent
* Have a diagnosis of RA per ACR criteria
* Must understand and voluntarily sign an informed consent form including writing consent for data protection
* Stable doses of methotrexate over the preceding 6 weeks

Exclusion Criteria:

* Pregnant or lactating females
* Previous anaphylactic response to vaccine components or to egg.
* Acute infection with T >38°C at the time of vaccination
* History of Guillain-Barre syndrome or demyelinating syndromes
* Previous vaccination with any live vaccine 4 weeks before or any inactivated vaccine 2 weeks before the study
* Blood transfusion within 6 months
* Active rheumatoid arthritis necessitating a recent change in the drug regimen
* Any other rheumatic disease such as systemic lupus erythematosus, mixed connective tissue disease, dermatomyositis/polymyositis, and vasculitis except for secondary Sjogren's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Doran MF, Crowson CS, Pond GR, O'Fallon WM, Gabriel SE. Frequency of infection in patients with rheumatoid arthritis compared with controls: a population-based study. Arthritis Rheum. 2002 Sep;46(9):2287-93. doi: 10.1002/art.10524. PMID 12355475
- [Background] McMahan ZH, Bingham CO 3rd. Effects of biological and non-biological immunomodulatory therapies on the immunogenicity of vaccines in patients with rheumatic diseases. Arthritis Res Ther. 2014 Dec 23;16(6):506. doi: 10.1186/s13075-014-0506-0. PMID 25587634
- [Background] Winthrop KL, Silverfield J, Racewicz A, Neal J, Lee EB, Hrycaj P, Gomez-Reino J, Soma K, Mebus C, Wilkinson B, Hodge J, Fan H, Wang T, Bingham CO 3rd. The effect of tofacitinib on pneumococcal and influenza vaccine responses in rheumatoid arthritis. Ann Rheum Dis. 2016 Apr;75(4):687-95. doi: 10.1136/annrheumdis-2014-207191. Epub 2015 Mar 20. PMID 25795907
- [Derived] Park JK, Lee MA, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Effect of methotrexate discontinuation on efficacy of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2017 Sep;76(9):1559-1565. doi: 10.1136/annrheumdis-2017-211128. Epub 2017 May 3. PMID 28468794

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Group 1 will continue MTX
  Methotrexate: Methotrexate will be continued
  Seasonal Influenza vaccine: all subjects will be vaccinated with a seasonal influenza vaccine
- Group 2: Group 2 will hold MTX 4 weeks before vaccination and resume MTX on the day of vaccination
  Methotrexate: Methotrexate will be continued
  Seasonal Influenza vaccine: all subjects will be vaccinated with a seasonal influenza vaccine
- Group 3: Group 3 will hold MTX 2 weeks before vaccination and resume MTX 2 weeks after vaccination
  Methotrexate: Methotrexate will be continued
  Seasonal Influenza vaccine: all subjects will be vaccinated with a seasonal influenza vaccine
- Group 4: Group 4 will hold MTX on day of vaccination and resume MTX 4 weeks after vaccination.
  Methotrexate: Methotrexate will be continued
  Seasonal Influenza vaccine: all subjects will be vaccinated with a seasonal influenza vaccine
Period: Visit 1- Visit 2
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 69 | 68 | 71 | 69
Completed | 59 | 49 | 57 | 63
Not Completed | 10 | 19 | 14 | 6
Period: Visit 2-Visit 3
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 59 | 49 | 57 | 63
Completed | 54 | 44 | 49 | 52
Not Completed | 5 | 5 | 8 | 11
Period: Visit 3- Visit 4
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 54 | 44 | 49 | 52
Completed | 53 | 43 | 47 | 50
Not Completed | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 54 | 44 | 49 | 52 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (13.1) | 58.5 (113.3) | 58.1 (10.9) | 58.1 (11.7) | 58.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 39 | 42 | 43 | 169
  Male | 9 | 5 | 7 | 9 | 30
Disease duration [Mean (Standard Deviation); unit: years] | 5.2 (4.5) | 6.1 (4.9) | 4.9 (4.4) | 6.2 (5.5) | 6.2 (5.5)
Disease Activity Score (DAS)-28 [Mean (Standard Deviation); unit: units on a scale (0-10)] — The Disease Activity Score (DAS) is a combined index to measure the disease activity in patients with Rheumatoid Arthritis (RA).
  The DAS will provide a number between 0 and 10, indicating how active the rheumatoid arthritis is at this moment, whereas a higher values represent a worse disease activity.
  0.. minimum score 10..maximum score
  units on a scale (0-10) | 2.5 (1.1) | 2.8 (1.2) | 2.6 (1.0) | 2.6 (1.0) | 2.6 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Satisfactory Vaccination Responses Against 3 Antigens
Description: Seroresponse is defined as serconversion or ≥4-fold increase in antibody titers
Time Frame: 8 weeks
Population: Per Protocol
Measure: Number; unit: percentage of responders
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
percentage of responders | 31.5 | 22.7 | 51 | 46.2

2. Secondary Outcome: Proportion of Seroprotection Against H1N1
Description: Seroprotection is defined as antibody titers of ≥40
Time Frame: 8 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 55 | 44 | 49 | 52
percentage of patients | 74 | 86 | 96 | 86

3. Secondary Outcome: Proportion of Seroprotection Against H3N2
Description: Seroprotection is defined as antibody titers of ≥40
Time Frame: 8 weeks
Measure: Number; unit: percentage of patients w/ seroprotection
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
percentage of patients w/ seroprotection | 100 | 96 | 98 | 96

4. Secondary Outcome: Proportion of Seroprotection Against B-Yamagata
Description: Seroprotection is defined as antibody titers of ≥40
Time Frame: 8 weeks
Measure: Number; unit: percentage of patients w/ seroprotection
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
percentage of patients w/ seroprotection | 72 | 71 | 94 | 81

5. Secondary Outcome: Change From Baseline in Antibody Titer Against H1N1
Description: Fold change = post-vaccination titer/pre-vaccination titer
Time Frame: Day of and 4 weeks after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
Fold change | 5.1 [3.4 to 7.8] | 5.0 [3.2 to 7.8] | 8.7 [5.3 to 14.5] | 8.1 [5.3 to 12.4]

6. Secondary Outcome: Change From Baseline in Antibody Titer Against H3N2
Description: Fold change = post-vaccination titer/pre-vaccination titer
Time Frame: Day of and 4 weeks after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
Fold change | 5.9 [4.3 to 8.1] | 6.1 [4.4 to 8.5] | 12.2 [8.4 to 17.5] | 10.0 [6.8 to 14.8]

7. Secondary Outcome: Change From Baseline in Antibody Titer Against B-Yamagata
Description: Fold change = post-vaccination titer/pre-vaccination titer
Time Frame: Day of and 4 weeks after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
Fold change | 2.9 [2.2 to 3.8] | 2.8 [2.1 to 3.7] | 4.7 [3.3 to 6.7] | 6.1 [4.2 to 8.8]

8. Secondary Outcome: DAS28 Flare Rate at Visit 4
Description: DAS28 flare rate at visit 4 as compared to visit 1. RA flare was defined as an increase in DAS28 of >1.2 (or >0.6 if the baseline DAS28 was ≥3.2).
Time Frame: 20 weeks from enrollment.
Measure: Number; unit: percentage of flare patients
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
percentage of flare patients | 7.5 | 14.0 | 19.1 | 12.0

9. Primary Outcome: Satisfactory Vaccination Responses Against > 2/3 Antigens
Description: Seroresponse is defined as serconversion or ≥4-fold increase in antibody titers
Time Frame: 8 weeks
Population: Per Protocol
Measure: Number; unit: percentage of responders
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
percentage of responders | 53.7 | 52.3 | 71.4 | 65.4

10. Primary Outcome: Satisfactory Vaccination Responses Against > 1/3 Antigens
Description: Seroresponse is defined as serconversion or ≥4-fold increase in antibody titers
Time Frame: 8 weeks
Population: Per Protocol
Measure: Number; unit: percentage of responders
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 44 | 49 | 52
percentage of responders | 77.8 | 81.8 | 87.8 | 88.5

ADVERSE EVENTS:
Time Frame: At each visit
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/54 | 2/44 | 0/49 | 0/52
Other Adverse Events (participants affected / at risk) | 33/54 | 23/44 | 23/49 | 17/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=54) | Group 2 (N=44) | Group 3 (N=49) | Group 4 (N=52)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=54) | Group 2 (N=44) | Group 3 (N=49) | Group 4 (N=52)
Upper respiratory infection (Infections and infestations) | 26 (26) | 18 (18) | 20 (20) | 16 (16)
Dizziness (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No